CLINICAL TRIAL: NCT02102685
Title: Vacuum Assisted Closure in Deep Neck Abscess
Brief Title: Vacuum Assisted Closure in Neck Abscess
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, CLOTILDE FUENTES OROZCO, PhD, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VACOTOL-012
Record Dates: First submitted 2014-03-27; First posted 2014-04-03 (Estimated); Last update posted 2014-04-22 (Estimated); Status verified 2014-04

CONDITIONS: Neck Abscess
Keywords: VAC Therapy; Neck Abscess; Traditional Therapy; Wound Healing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VAC Therapy (Active Comparator): active comparator: 14 patients within the first three days the VAC therapy was placed , proceeding as follows : organize the material , bandage removal , cleaning of the wound with irrigation solution , cut the sponge and placement on the wound , use of polyvinyl alcohol and / or silver foam, insertion of the tube seal and connection to the containing recipient.
  Interventions: Procedure: VAC Therapy
- Traditional Therapy (Placebo Comparator): 14 patients: after surgical drainage, a culture was taken, photographs every three days (during hospital stay ) and secretion culture; daily cleaning stipulated by the service was perform. The control of the patients were made until wound closure (presence of epithelialization tissue) .
  Interventions: Procedure: TRADITIONAL THERAPY

INTERVENTIONS:
Procedure: VAC Therapy — within the first three days the VAC therapy was placed , proceeding as follows : Wound cleaning was performed with irrigating solution and replacement of the sponges every 72 hours according to evolution, photographs were taken to assess the percentage of viable tissue and granulation. A Sample to culture was taken prior to placement of VAC therapy , during the use of it and at the time of removal of the system. When the wound presents clinical signs of improvement (elimination of purulent discharge and granulation tissue ) VAC therapy was withdrawn , and follow by delayed primary closure.
  Arms: VAC Therapy
Procedure: TRADITIONAL THERAPY — after surgical drainage, a culture was taken, photographs every three days (during hospital stay ) and secretion culture; daily cleaning stipulated by the service was perform. The control of the patients were made until wound closure (presence of epithelialization tissue) .
  Arms: Traditional Therapy

SUMMARY:
The presence of deep abscess in the neck is potentially severe, it can also lead to death in short term. The surgical treatment is indicated when there is commitment of the airway, critical condition, septicemia, complications, descendent infections, diabetes mellitus with no improving during the first 48 hours of parenteral antibiotic treatment and subsequent healing of the wounds until it heals by second intention. In this study investigators propose the use of vacuum Assisted Closure (VAC) that has been used satisfactorily to reduce edema, promote granulation, and ameliorate the tissue to afterwards reconstruct the defect, increase vascularity and diminish the bacterial load.

DETAILED DESCRIPTION:
Objective: To evaluate the therapeutic efficacy of the combination of vacuum-assisted in comparison with traditional therapy in wound healing in deep neck abscess.

Material and Methods Type of Study: Clinical Trial (Randomized) controlled This project was performed in patients from the Service of Otolaryngology, IMSS, diagnosed with deep neck abscess.

Procedure There were two groups: Group A, 14 patients treated with VAC therapy, group B, patients treated with conventional therapy Group A: within the first three days the VAC therapy will be placed , proceeding as follows : organize the material , bandage removal , cleaning of the wound with irrigation solution , cut the sponge and placement on the wound , use of polyvinyl alcohol and / or silver foam, insertion of the tube seal and connection to the containing recipient. Wound cleaning will performed with irrigating solution and replacement of the sponges every 72 hours according to evolution, photographs will be taken to assess the percentage of viable tissue and granulation. A Sample to culture will be taken prior to placement of VAC therapy , during the use of it and at the time of removal of the system. When the wound presents clinical signs of improvement (elimination of purulent discharge and granulation tissue ) VAC therapy will be withdrawn , and follow by delayed primary closure.

Patients will be assign to group B: 14 patients on admission, after surgical drainage, a culture will be taken, photographs every three days (during hospital stay ) and secretion culture; daily cleaning stipulated by the service will be perform. The control of the patients will be made until wound closure (presence of epithelialization tissue) .

Statistical Analysis Nominal variables will be analyzed using percentage frequencies, X2 test or Fisher exact test. Numeric variables using Student's t test for independent samples and ANOVA with post hoc Scheffe test. U Mann Whitney and Kruskal Wallis tests will be used as long as data do not conform to normal distribution. All values of p <0.05 will be considered statistically significant. The analysis will be perform with statistical program SPSS v. 18 for Windows program.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients of 18 years or older
* Diagnosis of Deep Neck Abscess users of the Mexican Institute of Social Security
* Incision from the anterior edge of the SCM muscle to unilateral or bilateral paratracheal line
* Spread of infection to a space larger than 7 cm
* Patients with systemic diseases

Exclusion Criteria:

* Patients with extensive necrosis of tissue that does not allow the suture of the wound
* Patients who for some reason do not conclude the study
* Patients with complications that require taking off the VAC Therapy
* Patients who miss their follow

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-09; Primary Completion 2011-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Granulation tissue percentage | every 3 days up to 3 months
  the percentage of granulation tissue will be evaluated by a software called image Image J

SECONDARY OUTCOMES:
complications | every 3 days up to 3 months
  haematoma, and wound dehiscence
microorganisms | every 7 days up to 3 months
  culture of the wound secretion

OTHER OUTCOMES:
mortality | Up to 6 months
  deaths registered during the study

CONTACTS AND LOCATIONS:
Overall Officials: Clotilde Fuentes-Orozco, PhD, Study Director — Instituto Mexicano del Seguro Social; Luis H Govea-Camacho, PhD, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Western Medical Center, Mexican Institute of Social Security, Guadalajara, Jalisco, Mexico